CLINICAL TRIAL: NCT06515522
Title: A Biological Signature for the Early Differential Diagnosis of Psychosis: Unveiling the Differences Between Mood Disorders and Schizophrenia With Multimodal Machine Learning Techniques
Brief Title: A Biological Signature for the Early Differential Diagnosis of Psychosis
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Francesco Benedetti, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PNRR-MCNT2-2023-12378015
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma and live cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schizophrenia: All patients with schizophrenia recruited from 2007 and 2023
  Interventions: Other: differential diagnosis
- Mood disorders: All patients with bipolar or major depressive disorders recruited from 2007 and 2023
  Interventions: Other: differential diagnosis
- Controls: healthy controls
  Interventions: Other: differential diagnosis

INTERVENTIONS:
Other: differential diagnosis — this is a retrospective observational study. no intervention has been or will be performed

SUMMARY:
Schizophrenia (SZ) and mood disorders (BD, MDD) are among the most disabling disorders worldwide, with a relevant social, functional, and economic burden. Although they are identified as distinct disorders, the potential overlapping symptomatology poses important challenges for the differential diagnosis. A consistent literature affirms that brain structure, and function reflect an intermediate phenotype of an underlying genetic vulnerability for the disorders, shaped by interaction with environmental experiences. Such experiences include early life stress and trauma which seem to characterize psychiatric patients and have been associated with brain abnormalities. Further, early life experiences have been associated with inflammation in a subpopulation of psychiatric patients However imaging, inflammatory, and genetic group-level differences, albeit consistent, do not impact clinical practice since they have not been translated into individual prediction. To address these issues, a rapidly growing body of scientific literature implemented computational techniques, such as machine learning (ML). In this project we will develop cutting-edge ML algorithms to predict the differential diagnosis between mood disorders and SZ from genetic, neuroimaging, inflammatory and environmental data in a unique cohort of 1850 patients and 1000 healthy controls recruited in 4 different centers in Italy. The project will address three different aims: in aim 1 we will develop algorithms for the differential diagnosis between SZ and MD combining multimodal neuroimaging and genetic data; in aim 2 we will predict the differential diagnosis between SZ and MD from immuno-inflammatory and environmental data; finally, with aim three we will exploit an animal model to identify the underlying mechanisms of brain alterations associated with exposure to early life stress. Machine learning analyses will include algorithms for data harmonization and feature reduction, as well as for generating normative models. Finally. different classifying models will be compared considering the specific features to achieve the best performance.The definition of reliable and objective biomarkers, combined with cutting-edge computational methodology, could help clinicians in providing more precise diagnoses and early interventions, also considering dimensional constructs & factors influencing outcomes such as affective vs non-affective psychosis and breadth of exposure to traumatic events

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65
2. diagnosed with Schizophrenia, Bipolar Disorder or Major depressive disorder.
3. For Bipolar and Major depressive disorder, Hamilton Depression Rating Scale scores >8
4. Multimodal 3 T MRI acquisition available (*)
5. Genetic and serum inflammatory data available, or serum and whole blood available for genotyping and inflammatory markers determination.

Exclusion Criteria:

1. Presence of major medical or neurological disorders
2. Alcohol or drugs abuse or dependence
3. Conditions known to alter immune-inflammatory status, such as rheumatic diseases, malignancies,
4. ongoing treatment with drugs acting on the immune system, such as corticosteroids, NSAIDs and other immunomodulatory drugs.
5. Pregnancy or lactating

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients with a diagnosis of Schizophrenia or Bipolar disorder or Major depressive disorder, neuroimaging data and peripheral blood sampling.
  Healthy controls with neuroimaging data and peripheral blood sampling
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Schizophrenia vs Mood disorders | baseline
  Predicting the differential diagnosis between Schizophrenia and Mood Disorders combining multimodal neuroimaging, immuno-inflammatory and genetic data

SECONDARY OUTCOMES:
Bipolar vs major depressive disorder | baseline
  Predicting the differential diagnosis between major depression and bipolar disorder, and the presence or absence of psychotic symptoms combining multimodal neuroimaging, immuno-inflammatory and genetic data

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Benedetti, Prof, Principal Investigator — IRCCS Ospedale San Raffaele